CLINICAL TRIAL: NCT02577575
Title: The Effects of Oxytocin on Social Cognition in Patients With Schizophrenia
Brief Title: Adult Oxytocin Study
Acronym: OT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joshua Woolley, Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10-01508
Record Dates: First submitted 2015-09-29; First posted 2015-10-16 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Schizophrenia; Oxytocin; Social Cognition
Keywords: Oxytocin; Syntocinon; Social Cognition; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): 40 IU Oxytocin
  Interventions: Drug: Oxytocin
- Saline Nasal Spray (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Saline Nasal Spray

INTERVENTIONS:
Drug: Oxytocin — 40 IU of the oxytocin will be administered intranasally for a one time dose at the beginning of the visit.
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Saline Nasal Spray — 40 IU of the saline nasal spray will be administered once at the beginning of the visit.
  Other Names: Placebo
  Arms: Saline Nasal Spray

SUMMARY:
In this study, investigators will examine the behavioral effects and neurophysiological mechanisms of the pro-social neuropeptide oxytocin in patients with recent-onset schizophrenia. Such research is a necessary first step towards identifying whether intranasal oxytocin administration can serve as an adjunct treatment for social impairments in schizophrenia.

Aim 1: To quantify the effects of exogenous oxytocin on social cognition and behavior in patients with recent-onset schizophrenia.

Hypothesis A: Patients and healthy comparison subjects will show enhanced social cognition (e.g., improved interpretation of paralinguistic and emotional cues, such as those involved in emotional or sarcastic communication) after administration of oxytocin versus placebo.

Hypothesis B: Patients and healthy comparison subjects will show increased attention to others' eyes and patients will exhibit increased facial affect expressivity after administration of oxytocin versus placebo.

Aim 2: To examine the effects of exogenous oxytocin on persistent negative symptoms in schizophrenia (PNS) activity in patients with recent-onset schizophrenia.

Hypothesis A: Patients and healthy comparison subjects will demonstrate increased PNS activity during social tasks after administration of oxytocin versus placebo.

Hypothesis B (exploratory): Patients and healthy comparison subjects' improvements in social cognition and behavior will be predicted by the degree to which oxytocin increases their PNS activity.

ELIGIBILITY:
Inclusion Criteria for Patients:

* 18 to 65 years of age
* English Speaking
* Meet Diagnostic and Statistical Manual (DSM)-IV criteria for schizophrenia, schizoaffective disorder, schizophreniform disorder.
* No or at most only minor changes to medications in the past week
* Able to use nasal spray
* Must be capable of providing informed consent

Inclusion Criteria for healthy volunteers:

* 18 to 65 years of age
* Clinically stable
* No diagnosis of mental disorder according to DSM-IV TR.
* Able to use nasal spray
* Must be capable of providing informed consent
* English Speaking

Exclusion Criteria:

* Active substance abuse or dependence as determined by a Urine Toxicology Drug Screening
* A current DSM-IV diagnosis of any disorder other than schizophrenia
* Medical conditions (atrophic rhinitis, recurrent nose bleeds and cranial-surgical procedures (hypophysectomy), congestion or sinus problems) that could interfere with the study as per the opinion of the investigator
* Hearing deficits
* Pregnancy
* Severe brain trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Improvement in social cognition task performance | 2-days at least 1-week apart
  The outcome will be the number of tasks that improve on the oxytocin day compared to the placebo day in a panel of tasks designed to measure the subject's level of social cognition. Participants will complete social cognition tasks, which include the Auction Task, Devil's Task, Ultimatum Task, Verbal Prosody, Effort Expenditure for Rewards Task (EEfRT), and Passive Viewing Eyetracking.

SECONDARY OUTCOMES:
Pre-morbid IQ Questionnaire (AmNART) | 1 day
  The American National Adult Reading Test (AMNART) is an instrument used to estimate premorbid verbal intelligence quotient (IQ) in adults. Participants are shown 45 words one at a time and are asked to read the word aloud. The scorer then writes 0 if the participant read the word incorrectly or 1 if the pronunciation is correct.
Experiences in Close Relationships-Relationship Structures (ECR-RS) Questionnaire | 1 day
  The ECR is used to evaluate the construct of adult attachment. The scale involves 36 itemized statements split into four parts, each part referring to a different attachment figure. Participants rank each item using a 7-point likert scale.
Childhood Trauma Questionnaire (CTQ) | 1 day
  The CTQ is a brief survey of 6 early traumatic experiences, including death, divorce, violence, sexual abuse, illness or other. The scale determines and assesses an individual's understanding of their childhood trauma, if applicable.
Emotional Quotient Scale (EQS) | 1 day
  The EQ is a 60-item self-report questionnaire that is designed to measure empathy in adults. Participants use a 4 item likert scale to record their responses (1=definitely agree, 4= definitely disagree).
Kinsey Scale | 1 day
  The Kinsey scale attempts to describe a person's sexual orientation using a scale from 0 (i.e. heterosexual) to 6 (i.e. homosexual).
Change in Working Memory capacity | 2-days at least 1-week apart
  This task determines a participant's working memory capacity using the University of Maryland Letter Number Span Assessment. This asks 24 questions of increasing working memory difficulty and the total correct is calculated. Investigators will measure the change in the total correct between oxytocin and placebo days.
Change in Auditory Perception correctness | 2-days at least 1-week apart
  The Sound Sweeps task determines auditory perception ability by measuring changes in pitches to sounds. Investigators will measure the change in the total correct responses between oxytocin and placebo days.
Change in Auditory Perception reaction time | 2-days at least 1-week apart
  The Sound Sweeps task determines auditory perception ability by measuring changes in pitches to sounds. Investigators will measure the change in the reaction time between oxytocin and placebo days.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Woolley, MD/PhD, Principal Investigator — University of California San Francisco, San Francisco Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California